CLINICAL TRIAL: NCT07044349
Title: Phase II Clinical Study of Utidelone Capsule (UTD2) in Patients With Advanced Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG02-2502
Record Dates: First submitted 2025-06-23; First posted 2025-06-30 (Actual); Last update posted 2025-06-30 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: UTD2; Utidelone Capsule
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Drug: Utidelone capsule 75mg/m2/d QD
- Cohort 2 initial group (Experimental)
  Interventions: Drug: Utidelone capsule 40mg/m2/d BID
- Cohort 2 escalation group (Experimental)
  Interventions: Drug: Utidelone capsule 50mg/m2/d BID
- Cohort 2 de-escalation group (Experimental)
  Interventions: Drug: Utidelone capsule 35mg/m2/d BID

INTERVENTIONS:
Drug: Utidelone capsule 75mg/m2/d QD — 75mg/m2/d, QD, D1-D5 for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: Cohort 1
Drug: Utidelone capsule 40mg/m2/d BID — 40mg/m2/d, BID, D1-D5 for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: Cohort 2 initial group
Drug: Utidelone capsule 50mg/m2/d BID — 50mg/m2/d, BID, D1-D5 for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: Cohort 2 escalation group
Drug: Utidelone capsule 35mg/m2/d BID — 35mg/m2/d, BID, D1-D5 for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: Cohort 2 de-escalation group

SUMMARY:
This is an open, multicenter, phase II clinical study enrolling patients with platinum-resistant advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer to evaluate the safety and efficacy of Utidelone Capsules. Approximately 72 patients will be included in this study.

DETAILED DESCRIPTION:
This study will be two cohorts:

Cohort 1: 30 participants are planned to be enrolled. The administration regimen is Utidelone Capsules at 75 mg/m2/d once a day. Fasting (fasting for 2 hours before administration and 1 hour after administration)is required from the 1st to the 5th day of each 21-day cycle.

Cohort 2: 6 to 12 participants are planned to be enrolled during the safety run-in part, and 30 participants are planned to be enrolled during the expansion part. The administration regimen is the twice daily (BID) administration of Utidelone capsules. The dosage of expansion part will be determined according to the safety run-in part. Fasting (fasting for 2 hours before administration and 1 hour after administration)is required from the 1st to the 5th day of each 21-day cycle.

The safety run-in part use a dose-escalation design. The initial dose was 40 mg/m2 of utidelone capsules BID. The escalation group was set at 50 mg/m2 BID or the de-escalation group at 35 mg/m2 BID. 6 participants will be enrolled in each dose group to evaluate dose-limiting toxicity (DLT).

After the completion of DLT observation during the safety run-in part, one administration regimen will be determined for the dose expansion period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who voluntarily sign the informed consent form, are willing and able to comply with the scheduled visits, study treatment plan, laboratory tests, and other study procedures.
2. Female participants aged ≥ 18 years when signing the informed consent form.
3. Pathologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal cancer.
4. Participants with at least one measurable lesion as defined per RECIST v1.1.
5. Participants must meet the criteria for platinum-resistant recurrence, which is defined as disease progression during platinum-based therapy or disease progression or recurrence within 6 months after the last platinum-based therapy. Note: Participants must have radiographically confirmed disease progression during or after the most recent line of systemic therapy. Biochemical progression is not considered disease progression in this study.
6. Participants must meet the requirements of failure or intolerance to the existing standard of treatment or no standard of treatment. Prior use of at least 1 but ≤ 3 lines of systemic antitumor treatment (neoadjuvant and adjuvant treatment are not considered prior systemic treatment, unless disease progression occurred during treatment or within 6 months after the last dose of treatment). Maintenance therapy (e.g., bevacizumab, poly-ADP ribose polymerase [PARP] inhibitors, hormonal therapy) is considered part of the prior line of treatment. Treatment changes due to toxicity without progression will be considered part of the prior line of treatment (i.e., not counted separately).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Hematology test within 7 days prior to enrollment (based on the laboratory normal range at each site), and no use of recombinant human granulocyte colony-stimulating factor (rhG-CSF) or blood products /erythropoietin (EPO) within 14 days prior to the laboratory test during the screening period.

   Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 100 × 109/L; Hemoglobin ≥ 9.0 g/dL.
9. Blood chemistry test within 7 days prior to enrollment (based on the laboratory normal range at each site); Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); ALT ≤ 3 × ULN (≤ 5 × ULN for participants with liver metastases); AST ≤ 3 × ULN (≤ 5 × ULN for participants with liver metastasis); Creatinine clearance (Ccr) ≥ 60 mL/min (calculated by Cockcroft-Gault formula).
10. Life expectancy ≥ 12 weeks.
11. Female participants of childbearing potential must agree to use highly effective contraceptive methods and not to donate eggs during the study and for 8 weeks after the last dose of study treatment. Female patients of childbearing potential must have a negative blood or urine pregnancy test result at screening and be willing to undergo additional pregnancy tests as needed throughout the study. See Appendix 1 for details.

Exclusion Criteria:

1. The best overall response during the first-line platinum-based treatment is disease progression, or disease recurrence or progression within 3 months after the end of the platinum-based treatment.
2. History of other malignancies within 5 years prior to enrollment, excluding cured skin basal cell carcinoma, cervical carcinoma in situ, or papillary thyroid carcinoma.
3. Anti-tumor therapy, including chemotherapy, radiotherapy, target therapy, immunotherapy, etc. within 4 weeks prior to the first dose of the investigational drug, except for the following items;

   1. Received nitrosourea or mitomycin C within 6 weeks prior to the first dose of the investigational drug;
   2. Oral fluorouracil, small molecule targeted drugs, or endocrine therapy within 2 weeks or within 5 half-lives of the drug prior to the first dose of the investigational drug, whichever is shorter;
   3. Use of traditional Chinese medicine with anti-tumor indications or endocrine therapy within 2 weeks prior to the first dose of the investigational drug.
4. Participants who have undergone major surgery (craniotomy, thoracotomy, or laparotomy, or as defined by the investigator) or have experienced significant trauma within 4 weeks prior to the first dose of the investigational product, or those who require elective surgery during the study.
5. Participants with adverse reactions due to previous antitumor therapy that have not recovered to Grade ≤1 (based on CTCAE 5.0), except toxicities without safety risks as judged by the investigator, such as alopecia.
6. Participants with gastrointestinal perforation, gastrointestinal fistula, or intra-abdominal abscess, or patients with gastrointestinal hemorrhage, gastrointestinal obstruction (including paralytic ileus), or imaging/clinical symptoms suggestive of bowel obstruction within 3 months prior to the first use of the investigational product;
7. Participants who are unable to take oral medications, or with other factors that interfere with the oral administration and absorption of the drug, or those who require total parenteral nutrition.
8. Participants who need concomitant use of strong CYP3A4 inhibitors or inducers, or medications that prolong the QT interval, within 14 days prior to the first use of the investigational product or during the study.
9. Participants with symptomatic or uncontrolled central nervous system (CNS) metastases or meningeal metastases, i.e., patients with brain metastasis disease progression confirmed by examination within 2 months after radiotherapy or other local treatments, or patients who are judged by the investigator to be unsuitable for enrollment.
10. Uncontrolled bone metastases, i.e., patients who have experienced fracture or have the risk of fracture in recent days, patients who need surgery or localized radiotherapy in recent days, or those with other critical conditions as determined by the investigator.
11. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once per month or more frequently).
12. History of severe cardiovascular and cerebrovascular diseases, including but not limited to:

    Patients with acute myocardial infarction, severe/uncontrolled angina, or coronary artery bypass surgery within 6 months prior to the first dose of the investigational product; congestive heart failure with a New York Heart Association (NYHA) classification ≥ 2; left ventricular ejection fraction (LVEF) < 50%; Fridericia corrected QT interval > 470 ms (average of three measurements); or a history of myocarditis (including patients with a past history of myocarditis that recovered after treatment) or other Grade ≥ 3 cardiovascular events.

    Stroke and/or transient ischemic attack within 6 months prior to the first dose of the investigational product; Uncontrolled hypertension despite standard treatment; Other heart diseases at high risk, as judged by the investigator.
13. Participants with uncontrolled diabetes mellitus.
14. Participants with active hepatitis B and/or hepatitis C, i.e., HBsAg positive and HBV DNA positive; anti-HCV positive and HCV RNA positive; positive for human immunodeficiency virus (HIV) antibody; positive for treponema pallidum specific antibody.
15. Participants who had active infection prior to screening and initial use of the investigational drug and required systemic anti-infective therapy.
16. Pregnant or breastfeeding women, or women who plan to become pregnant during the study.
17. Participants with mental disorder or poor compliance.
18. Participants with prior use of utidelone.
19. Participants with known hypersensitivity to the investigational product or any of the excipients.
20. Participants who simultaneously participate in another interventional clinical trial or use other investigational therapies.
21. Participants who, in the opinion of the investigator, are not suitable to participate in this study due to history of severe systemic diseases or other reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and the maximum tolerated dose of the BID administration regimen | Until 21 days after the first dose of treatment
The incidence of adverse events (AE)/serious adverse events (SAE) | Until 28 days after the last dose of treatment

SECONDARY OUTCOMES:
Objective response rate (ORR) | 18 months
  based on RECIST v1.1
Disease control rate (DCR) | 18 months
Progression-free survival (PFS) | 18 months
Maximum (or peak) serum concentration-Cmax | 18 months
Time to peak drug concentration-Tmax | 18 months
The area under the concentration-time curve from dosing (time 0) to time t-AUC0-t | 18 months
The time required for plasma concentration of a drug to decrease by 50%-t1/2 | 18 months

IPD SHARING:
Plan to Share IPD: No